CLINICAL TRIAL: NCT04849403
Title: EVALUATION OF THE FREQUENCY OF TROCAR SITE HERNIA AFTER LAPAROSCOPIC SLEEVE GASTRECTOMY
Brief Title: TROCAR SITE HERNIA AFTER LSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, MD. Anil Ergin, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DR.ANIL ERGIN
Record Dates: First submitted 2021-04-10; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Obesity, Morbid; Hernia Incisional
Keywords: Laparoscopic Sleeve Gastrectomy; Morbid obesity; Trocar site hernia; Carter Thomasson Suture Passer
MeSH Terms: conditions — Obesity, Morbid; Incisional Hernia

STUDY DESIGN:
Intervention Model Description: 61 patients who underwent Laparoscopic Sleeve Gastrectomy are included. USG was performed (Figure I,II) by a clinician who had previously received superficial USG evaluation training for trocar site hernia and abdominal incision sites were investigated for the presence of hernias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The group USG was applied (Other): USG was applied to the patients who underwent Laparoscopic sleeve gastrectomy for research trocar site hernia after 2-4 years from the surgery. Carter Thomasson suture passer was used to close fascial defect in all patients.
  Interventions: Procedure: CTSP

INTERVENTIONS:
Procedure: CTSP — In all patients Carter Thomasson Suture Passer (CTSP) were used for closing fascial defect peroperatively

SUMMARY:
Today, laparoscopic sleeve gastrectomy (LSG) has become the most frequently performed bariatric surgical method. One of the complications seen after LSG is trocar site hernia (TSH). There is no clear information about the rate of TSH detected radiologically after LSG. Thick abdominal wall and failure to adequately expose the facial defect related to this, mobility limitations due to excessive subcutaneous fatty tissue are the reasons accused for increased incidence of TSH.

Demographic characteristics and postoperative weight loss of patients who underwent LSG procedure in our clinic between January 2015 and June 2017 and whose facial defects in the trocar region were repaired with the Carter-Thomason Suture Passer (CTSP) were evaluated. TSH evaluation was made both by physical examination and superficial USG by a general surgeon who had radiological training on concurrent superficial abdominal ultrasonography (USG). Detected TSHs were divided into two groups as symptomatic and asymptomatic.

DETAILED DESCRIPTION:
This study included 61 patients who applied to the obesity follow-up outpatient clinic for any complaints or routine control over a 3-month period or who were called by telephone for control and who underwent laparoscopic sleeve gastrectomy for morbid obesity between January 2015- June 2017. Patients with symptoms associated with trocar site hernia were also included in the study, while patients with multiple bariatric surgical procedures or abdominal operations were excluded. Physical examinations to detect hernias were performed both in standing and supine positions for all patients and also during increased abdominal pressure by the Valsalva maneuver. All abdominal incision sites were examined. On physical examination, a hernia was defined as a bulging during the Valsalva maneuver and palpation of the fascial defect. USG was performed (Figure I,II) by a clinician who had previously received superficial USG evaluation training for trocar site hernia with a GE pro 500, 3 MHz and abdominal incision sites were investigated for the presence of hernias.

The trocar entry localizations of the patients were all the same and are as follows: one 15-mm camera trocar (supraumbilical) , one 10-mm working trocar (left upper quadrant), two 5-mm working trocars (right and left upper quadrant) and one 5-mm liver retractor. Trocar entry localizations are shown in Figure III. During fascia closure procedure, No. 0 absorbable suture (PolyglactinYü-ce Vicryl Ⓡ, Tekirdag, Turkey ) was used with the CTSP (Figure IV). The collected data were recorded in a pre-established database with age, gender, Diabetes Mellitus (DM), postoperative follow-up period, BMI at the time of operation and BMI during superficial USG.

This study was approved by the Ethics Committee of University of Health Sciences Istanbul Fatih Sultan Mehmet Training and Research Hospital (12.09.2019 / 80).

ELIGIBILITY:
Inclusion Criteria:

* The patients above 18 years old.
* The patient who went Laparoscopic Sleeve Gastrectomy (LSG) procedure for morbid obesity.

Exclusion Criteria:

* The patients who needed to have additional surgery after the LSG in their follow up.
* The patients who could not reached and did not attend to the Ultrasound examination.
* The patient who did not approve the participate to the study.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
incidence of incisional hernia | 2-4 years
  Superficial abdominal Ultrasound for the incisional hernia to trocar sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Anıl Ergin, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided